CLINICAL TRIAL: NCT07275164
Title: Revolutionizing Musculoskeletal Shoulder Pain Management: High-intensity Interval Training as a Systemic Intervention. A Feasibility Study.
Brief Title: HIIT for Inflammatory-driven Shoulder Pain.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Michel GCAM Mertens, Dr., Universiteit Antwerpen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 7796
Record Dates: First submitted 2025-11-17; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Chronic Shoulder Pain; Rotator Cuff Related Shoulder Pain; Frozen Shoulder; Shoulder Adhesive Capsulitis; Shoulder Pain
Keywords: low-grade inflammation; chronic shoulder pain; autonomic dysfunction; metabolic syndrome; frozen shoulder; rotator cuff related shoulder pain; high intensity interval training
MeSH Terms: conditions — Bursitis; Shoulder Pain; Primary Dysautonomias; Metabolic Syndrome | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Only the group with shoulder pain will receive one intervention session. The asymptomatic controls are recruited for comparing baseline values.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High intensity interval training (HIIT) (Experimental): One 20-minute HIIT session (5x1 min at VO₂max with 1 min recovery at 50% VO₂max) on cycle ergometer
  Interventions: Other: High intensity interval training (HIIT)

INTERVENTIONS:
Other: High intensity interval training (HIIT) — One 20-minute HIIT session (5x1 min at VO₂max with 1 min recovery at 50% VO₂max) on cycle ergometer.

SUMMARY:
This feasibility study investigates whether high-intensity interval training (HIIT) is feasible and acceptable for individuals with long-term shoulder pain where low-grade inflammation is suspected. Many patients do not recover fully with current local treatments, and systemic factors such as inflammation, and metabolic changes, additionally disturbances in the functioning of the nervous system often seem to play a role. HIIT is a time-efficient form of exercise that has been shown to improve inflammation and metabolic values and positively influence the balance of the nervous system. In this feasibility study, the investigators are enrolling 15 individuals with persistent shoulder pain (diagnosed with rotator cuff-related shoulder pain or frozen shoulder) with >3 months of symptoms, and 15 individuals without shoulder complaints. All participants will undergo measurements of inflammatory levels, glycosylated hemoglobin (HbA1c), blood pressure, body composition, pain sensitivity tests, and complete questionnaires about autonomic complaints and quality of life. Participants with shoulder pain will also perform one personalized HIIT session on a cycle ergometer. The investigators will assess whether participants accept a systemic intervention for their shoulder pain, if they are cooperative, and how they feel about the session; additionally, any side effects will be recorded. The aim is to determine whether HIIT is practically feasible and safe for this group and whether there are indications that systemic factors such as inflammation and nervous system function are associated with persistent shoulder pain. The outcome will determine whether follow-up research with a larger study is worthwhile.

DETAILED DESCRIPTION:
Persistent musculoskeletal shoulder pain, such as rotator cuff-related complaints and frozen shoulder, is common and often leads to long-term limitations and reduced quality of life. Despite available treatment options, including exercise therapy, manual techniques and infiltrations, a significant group of patients do not experience full recovery. Growing scientific evidence suggests that chronic low-grade inflammation, metabolic disorders, such as insulin resistance or obesity, autonomic dysfunction, and changes in somatosensory processing contribute to the persistence of complaints. Within this framework, physical activity is receiving more attention as a systemic intervention. High-intensity interval training (HIIT) in particular appears to have a pronounced effect on inflammatory levels, metabolic parameters, cardiovascular function, and pain modulation in various populations. HIIT also offers practical advantages due to its short duration and higher efficiency compared to traditional endurance training. Therefore, the primary aim of the current study is to investigate the feasibility of a HIIT protocol in individuals with chronic inflammatory-driven shoulder pain. This investigation includes recruitment rate, adherence, acceptance, satisfaction, motivation, safety, and practical feasibility. A secondary aim of the current study is to explore differences between individuals with shoulder pain and asymptomatic controls in terms of inflammatory markers (C-Reactive Protein), metabolic parameters (HbA1c, blood pressure, body composition), autonomic functions (self-reported symptoms, heart rate variability) and somatosensory functions (pressure pain thresholds, temporal summation and conditioned pain modulation). This is a cross-sectional feasibility study with 30 participants (15 individuals with chronic shoulder pain and 15 asymptomatic controls). The individuals with shoulder pain participate in two sessions: a maximal exercise test on a cycle ergometer (to determine VO₂max and Wmax) and a combined assessment and HIIT session. Asymptomatic controls undergo a single assessment session. The HIIT protocol consists of five one-minute intervals of cycling at 100% of the individually determined VO₂max capacity, alternating with one minute of active rest at 50% of this capacity. The total exercise time is approximately 20 minutes. The session is supervised by an experienced physiotherapist in a research setting (MOVANT, University of Antwerp). Clinical parameters that will be assessed and stored in REDCap include demographics, shoulder pain and disability (SPADI), pain intensity (VAS), quality of life (EQ-5D), inflammation (c-reactive protein), nutrition-related inflammatory index, metabolic markers (glycosylated hemoglobin, blood pressure and body composition through bioelectrical impedance), autonomic functions (self-reported autonomic symptoms and Heart Rate Variability), and somatosensory processing (pressure pain thresholds, temporal summation, and conditioned pain modulation). Results are mainly reported descriptively, with confidence intervals to estimate effect sizes. As this is a pilot study, the design is not powered for formal hypothesis testing.The study aims to investigate whether HIIT is feasible and safe in this population and to provide initial indications of the role of systemic processes in the persistence of shoulder complaints. The results may form the basis for larger randomized studies and may contribute to a paradigm shift towards systemic approaches in the treatment of musculoskeletal pain.

ELIGIBILITY:
Inclusion Criteria:

Shoulder pain group

* Shoulder pain > 3 months
* Diagnosis of rotator cuff related shoulder pain or frozen shoulder
* Understanding Dutch in speaking and writing.

Control group

o Understanding Dutch in speaking and writing

Exclusion Criteria:

Shoulder pain group

* <18 years
* Shoulder surgery or trauma in past year
* Neurological, cancer, or neuromuscular disease
* Osteoarthritis, cervical or AC joint pathology
* Heavy physical exertion <48h before testing

Control group

* <18 years
* recent or recurrent neck/shoulder pain
* systemic or neurological disease
* psychiatric disorders
* pregnancy/breastfeeding
* pain medication <48h before test

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Participant acceptance and satisfaction | Immediately after the HIIT training session
  Participant acceptance and satisfaction of the HIIT-session will be assessed with an adapted short questionnaire based on the total shoulder arthroplasty postoperative satisfaction questionnaire.
HIIT protocol adherence | During the training session
  HIIT protocol adherence will be assessed by determining the percentage of HIIT-protocol completers and registration of protocol adjustments.
Intrinsic motivation | Immediately after the training session
  Intrinsic motivation of the participants with shoulder pain will be assessed using the intrinsic motivation inventory (IMI). From this questionnaire only the following domains will be questioned: interest/enjoyment, effort, and value/usefulness. The questions will be adapted specific to the current study, as recommended.
Study recruitment rate | During the study period
  Study recruitment rate will be determined by dividing the number of participants by the number of contacted individuals. Reasons for non-participation will be assessed with preset response options.
Full protocol conduction | Immediately after the assessment and training session
  Assessment of full protocol conduction will be assessed by registering preparation time, protocol duration, and issues with equipment and location.
Adverse events | Up to 3 days after training and assessment
  The severity of the adverse event will be determine based on the Common Terminology Criteria for Adverse Events (CTCAE).

SECONDARY OUTCOMES:
Shoulder pain and disability | Baseline
  The shoulder pain and disability index (SPADI) will be used, this is a self-reported index that consists of 13 items in two domains (pain (5 items) and disability (8 items)). A percentage ranging from 0 (no pain or disability) to 100 (worst pain or disability) will be used to present the pain and disability experienced by the participants. The SPADI has been found valid and reliable in evaluating pain and disability in shoulder disorders.
Pain intensity | Baseline
  Pain intensity will be measured by a visual analogue scale. Participants will be asked to rate their pain on a 10 cm line by drawing a vertical mark on that line. The left end of the line represents 'No pain' (0 cm) and the right end 'Most severe pain' (10 cm). The scoring is the distance (in millimeter) from the left end of the line to the vertical mark of the participant. Participants must rate their shoulder pain for three moments: current and minimal and maximal pain during the last week. The VAS has been found valid and reliable.
Health-related quality of life | Baseline
  Health-related quality of life will be assessed with the EQ-5D. The EQ-5D is a standardized, validated measure comprising five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is rated on a five-level ordinal scale (from 'no problems' to 'extreme problems'), offering improved sensitivity and reduced ceiling effects compared to the earlier 3-level version. Additionally, the EQ-5D includes a visual analogue scale (EQ-VAS), on which participants rate their overall health on a scale ranging from 0 ("the worst health you can imagine") to 100 ("the best health you can imagine"). The psychometric properties of the EQ-5D are excellent in a broad range of populations, conditions and settings. Utility scores will be calculated using the Dutch EQ-5D value set.
C-reactive protein level | Baseline
  C-reactive protein (CRP) level will be measured by the QuikRead go easy CRP, a highly sensitive tool. With 10 μL blood (fingerprick) the level of CRP between 1 and 120 mg/L can be determined within 5 minutes. This tool has been found reliable.
Adapted dietary inflammatory index | Baseline
  The adapted dietary inflammatory index (ADII) will be based on data acquired through the food frequency questionnaire (FFQ), as conducted previously. The ADII is a literature-derived index that summarizes an individual's diet on the continuum from maximally anti-inflammatory to maximally pro-inflammatory. ADII was calculated by multiplying the dietary inflammatory weights of the dietary components by the daily intake.
Glycosylated hemoglobin | Baseline
  Glycosylated hemoglobin (HbA1c) will be measured with the A1CNOW+ tool. The A1CNOW+ is a tool that measures the A1c and total hemoglobin and determines the percentage HbA1c over the last 90 days, which is valid and reliable.
Blood pressure | Baseline
  Blood pressure will be measured using an automated office blood pressure monitor in a seated position in a quit examination room. Both diastolic and systolic pressure will be recorded.
Body composition | Baseline
  Body composition will be determined by the InBody 770® (InBodyUSA, Cerritos, CA), more specifically %body fat and fat free mass of the participants will be determined.
Self-reported autonomic symptoms | Baseline
  Self-reported autonomic symptoms will be assessed by the composite autonomic symptom score 31 (COMPASS-31), which has 31 questions in six domains (orthostatic intolerance, vasomotor, secretomotor, gastrointestinal, constipation, bladder, and pupillomotor). Total score ranges from 0 to 100 because of summation of the six subdomains.
Vasomotor function | Baseline
  Vasomotor function of the autonomic nervous system (parasympathetic branch) will be measured with the help of resting heart rate variability (HRV), which will be measured using a chest strap (polar H10). The root mean square of successive RR-interval differences (RRSMD), mean RR interval, standard deviation of all normal RR intervals (SDNN), and percentage of successive RR intervals that differ by more than 50 ms (pNN50) will be determined.
Primary and secondary hyperalgesia | Baseline
  Primary and secondary hyperalgesia (in kg/cm2) will be assessed by pressure pain thresholds (PPTs). The PPTs will be determined at both affected and unaffected (shoulder pain group) and dominant and non-dominant (control group) shoulders and affected side (shoulder pain group) or dominant (control group) quadriceps muscle.
Temporal summation | Baseline
  Temporal summation will be induced with a train of 10 repeated pressure stimuli at the quadriceps muscle at the affected (shoulder pain group) or dominant (control group) side using a digital algometer. Pressure will be applied with 2 kg/s with 1-second interstimulus intervals. The pressure for temporal summation will be the mean PPT previously determined for the quadriceps. Participants rate their pain intensity on a NRS (0-10) after the first, fifth, and tenth repetition of the train stimuli. Temporal summation is calculated as the difference in pain intensity between the tenth and the first pulse
Conditioned pain modulation | Baseline
  The test stimulus consists of mechanical pressure pain elicited (PPT). The conditioning stimulus consists of ischemic occlusion and will be applied to the unaffected (shoulder pain group) or non-dominant (control group) arm with an inflatable air cuff (Boso Profitest). The absolute conditioned pain modulation effect will be calculated as the difference between the PPT at baseline and the PPT with conditioning stimulus, while the relative effect will be calculated as follows: (PPT at baseline - PPT with conditioning stimulus) / PPT at baseline.

OTHER OUTCOMES:
Gender | Baseline
  The gender of the participant
Age | Baseline
  The age of the participant
Job status | Baseline
  The job status of the participant
Alcohol abuse | Baseline
  The alcohol abuse status of the participant
Smoking status | Baseline
  Smoking status of the participant
Comorbidities | Baseline
  Presence and type(s) of comorbidities of the participant
Disorder characteristics | Baseline
  Characteristics of the disorder the participant presents with

CONTACTS AND LOCATIONS:
Overall Officials: Michel Mertens, PhD, Principal Investigator — Universiteit Antwerpen
Locations (1):
- Universiteit Antwerpen, Wilrijk, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The results of the food frequency questionnaire, which is part of the nutritional inflammatory index, will be shared with the developers of the questionnaire for optimization of the questionnaire. Furthermore, all data can be shared with other researchers upon reasonable request. Data will not be publicly available.
Time Frame: It will only be available upon reasonable request.
Access Criteria: The requested data will be send to the requester by the PI of the study and a data sharing agreement will be signed by both parties.